CLINICAL TRIAL: NCT03668860
Title: A Phase 1, Open-Label, Randomized Study to Compare the Pharmacokinetics and Pharmacodynamics of Single Dose Dexamethasone and Betamethasone Administered Orally and Intramuscularly in Healthy Female Subjects
Brief Title: India Dexamethasone and Betamethasone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Syngene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIN001 - India Steroids
Record Dates: First submitted 2018-08-10; First posted 2018-09-13 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Preterm Birth; Antenatal Corticosteroids
Keywords: Antenatal Corticosteroids; Betamethasone; Dexamethasone
MeSH Terms: conditions — Premature Birth | interventions — Dexamethasone; Betamethasone; betamethasone acetate phosphate; Suspensions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Treatments A & B (6 subjects) (Active Comparator): After overnight fasting of at least 10 hours, a single dose of investigational product A will be administered intramuscularly at gluteal or thigh region to each subject in this arm.
  Following washout period of between 9-12 days and after overnight fasting of at least 10 hours, a single dose of investigational product B will be administered intramuscularly at gluteal or thigh region to each subject in this arm.
  (Treatment A: Dexamethasone sodium phosphate intramuscular injection, 4mg/mL - Total dose: 1.5mL (6mg))
  (Treatment B: Betamethasone phosphate solution intramuscular injection, 4mg/mL - Total dose: 1.5mL (6mg))
  Interventions: Drug: Dexamethasone 4 mg/ml; Drug: Betamethasone 4 mg/ml
- Treatments B & A (6 subjects) (Active Comparator): After overnight fasting of at least 10 hours, a single dose of investigational product B will be administered intramuscularly at gluteal or thigh region to each subject in this arm.
  Following washout period of between 9-12 days and after overnight fasting of at least 10 hours, a single dose of investigational product A will be administered intramuscularly at gluteal or thigh region to each subject in this arm.
  (Treatment B: Betamethasone phosphate solution intramuscular injection, 4mg/mL - Total dose: 1.5mL (6mg))
  (Treatment A: Dexamethasone sodium phosphate intramuscular injection, 4mg/mL - Total dose: 1.5mL (6mg))
  Interventions: Drug: Dexamethasone 4 mg/ml; Drug: Betamethasone 4 mg/ml
- Treatments C & D (6 subjects) (Active Comparator): After overnight fasting of at least 10 hours, a single dose of investigational product C will be administered intramuscularly at gluteal or thigh region to each subject in this arm.
  Following washout period of between 9-12 days and after overnight fasting of at least 10 hours, a single dose of investigational product D will be administered orally with 240± 2mL of water in sitting posture at room temperature to each subject in this arm.
  (Treatment C: Celestone Soluspan intramuscular injection, 6mg/mL (3mg phosphate and 3 mg acetate salts) - Total dose: 1mL (6mg))
  (Treatment D: Dexamethasone phosphate 0.5mg oral tablets - Total dose: 12 tablets (6mg))
  Interventions: Drug: Celestone Soluspan 6Mg/Ml Suspension for Injection; Drug: Dexamethasone Oral Tablet
- Treatments D & C (6 subjects) (Active Comparator): After overnight fasting of at least 10 hours, a single dose of investigational product D will be administered orally with 240± 2mL of water in sitting posture at room temperature to each subject in this arm.
  Following washout period of between 9-12 days and after overnight fasting of at least 10 hours, a single dose of investigational product C will be administered intramuscularly at gluteal or thigh region to each subject in this arm.
  (Treatment D: Dexamethasone phosphate 0.5mg oral tablets - Total dose: 12 tablets (6mg))
  (Treatment C: Celestone Soluspan intramuscular injection, 6mg/mL (3mg phosphate and 3 mg acetate salts) - Total dose 1mL (6mg))
  Interventions: Drug: Celestone Soluspan 6Mg/Ml Suspension for Injection; Drug: Dexamethasone Oral Tablet
- Treatments E & D (6 subjects) (Active Comparator): After overnight fasting of at least 10 hours, a single dose of investigational product E will be administered orally with 240± 2mL of water in sitting posture at room temperature to each subject in this arm.
  Following washout period of between 9-12 days and after overnight fasting of at least 10 hours, a single dose of investigational product D will be administered orally with 240± 2mL of water in sitting posture at room temperature to each subject in this arm.
  (Treatment E: Betamethasone phosphate 0.5mg oral tablets - Total dose: 12 tablets (6mg))
  (Treatment D: Dexamethasone phosphate 0.5mg oral tablets - Total dose: 12 tablets (6mg))
  Interventions: Drug: Dexamethasone Oral Tablet; Drug: Betamethasone Oral Tablet
- Treatments D & E (6 subjects) (Active Comparator): After overnight fasting of at least 10 hours, a single dose of investigational product D will be administered orally with 240± 2mL of water in sitting posture at room temperature to each subject in this arm.
  Following washout period of between 9-12 days and after overnight fasting of at least 10 hours, a single dose of investigational product E will be administered orally with 240± 2mL of water in sitting posture at room temperature to each subject in this arm.
  (Treatment D: Dexamethasone phosphate 0.5mg oral tablets - Total dose: 12 tablets (6mg))
  (Treatment E: Betamethasone phosphate 0.5mg oral tablets - Total dose: 12 tablets (6mg))
  Interventions: Drug: Dexamethasone Oral Tablet; Drug: Betamethasone Oral Tablet
- Treatments C & E (6 subjects) (Active Comparator): After overnight fasting of at least 10 hours, a single dose of investigational product C will be administered intramuscularly at gluteal or thigh region to each subject in this arm.
  Following washout period of between 9-12 days and after overnight fasting of at least 10 hours, a single dose of investigational product E will be administered orally with 240± 2mL of water in sitting posture at room temperature to each subject in this arm.
  C: Celestone Soluspan intramuscular injection, 6mg/mL (3mg phosphate and 3 mg acetate salts) - Total dose 1mL (6mg)
  E: Betamethasone phosphate 0.5mg oral tablets - Total dose: 12 tablets (6mg)
  Interventions: Drug: Celestone Soluspan 6Mg/Ml Suspension for Injection; Drug: Betamethasone Oral Tablet
- Treatments E & C (6 subjects) (Active Comparator): After overnight fasting of at least 10 hours, a single dose of investigational product E will be administered orally with 240± 2mL of water in sitting posture at room temperature to each subject in this arm.
  Following washout period of between 9-12 days and after overnight fasting of at least 10 hours, a single dose of investigational product C will be administered intramuscularly at gluteal or thigh region to each subject in this arm.
  E: Betamethasone phosphate 0.5mg oral tablets - Total dose: 12 tablets (6mg)
  C: Celestone Soluspan intramuscular injection, 6mg/mL (3mg phosphate and 3 mg acetate salts) - Total dose 1mL (6mg)
  Interventions: Drug: Celestone Soluspan 6Mg/Ml Suspension for Injection; Drug: Betamethasone Oral Tablet

INTERVENTIONS:
Drug: Dexamethasone 4 mg/ml — Intramuscular. Total dose: 1.5 mL (6 mg)
  Arms: Treatments A & B (6 subjects); Treatments B & A (6 subjects)
Drug: Betamethasone 4 mg/ml — Intramuscular. Total dose: 1.5 mL (6 mg)
  Arms: Treatments A & B (6 subjects); Treatments B & A (6 subjects)
Drug: Celestone Soluspan 6Mg/Ml Suspension for Injection — Intramuscular. Total dose: 1 mL (6 mg)
  Arms: Treatments C & D (6 subjects); Treatments C & E (6 subjects); Treatments D & C (6 subjects); Treatments E & C (6 subjects)
Drug: Dexamethasone Oral Tablet — Oral. Total dose: 12 Tablets (6 mg)
  Arms: Treatments C & D (6 subjects); Treatments D & C (6 subjects); Treatments D & E (6 subjects); Treatments E & D (6 subjects)
Drug: Betamethasone Oral Tablet — Oral. Total dose: 12 Tablets (6 mg)
  Arms: Treatments C & E (6 subjects); Treatments D & E (6 subjects); Treatments E & C (6 subjects); Treatments E & D (6 subjects)

SUMMARY:
An open label, randomized, two-period, crossover, study to compare the pharmacokinetics and pharmacodynamics of single dose Dexamethasone and Betamethasone administered orally and intramuscularly in 48 healthy, adult, female subjects under fasting conditions. This study is being conducted in Bangalore, India.

ELIGIBILITY:
Inclusion Criteria:

1. - Healthy, adult, female subjects within the age range of 18 to 40 years [both inclusive].
2. - Weight not less than 45 kg.
3. - BMI [18.00 to 25.00 kg/m2] [both inclusive].
4. - Willingness to provide written informed consent to participate in the study.
5. - Without any medical or surgical condition that might interfere with gastrointestinal absorption of the study drug.
6. - Free of significant diseases or clinically significant abnormal findings during screening, medical history, physical examination, laboratory evaluations, 12-lead ECG, Chest X-ray [PA view].
7. - Subjects should be non-smoker or moderate smokers (less than 10 cigarettes a day), and should not be consuming tobacco containing products [ defined as someone who has stopped smoking for a year from the date of screening].
8. - Subject must be either a non-drinker or an occasional drinker of alcohol and agreed to abstain from alcoholic consumption during the study duration.
9. - Absence of disease markers of HIV I and 2, Hepatitis Band C and Syphilis.
10. - Female subjects of childbearing potential must be using two acceptable methods of contraception, ( e.g., intra-uterine device (IUD) plus condom, spermicidal gel plus condom, diaphragm plus condom, progestin only implants and long acting injectables (Depo Provera), etc.). These measures are required during the study and for at least two weeks after the last dose and conveyed during the inform consent process (or) postmenopausal women for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy have been performed).
11. - Subject should be literate.

Exclusion Criteria:

1. - History or presence of significant: Cardiovascular, pulmonary, hepatic, renal, hematological, gastro- intestinal, endocrine, immunologic, dermatologic, neurological, HEENT (Head, Eyes, Ears, Nose And Throat), psychiatric disease/ disorder.
2. - History or presence of significant:

   * Asthma, urticaria or other allergic type reactions or hypersensitivity after taking Dexamethasone or Betamethasone or any other drug.
   * Ulceration or history of gastric and / or duodenal ulcer.
   * Stomach or intestinal bleeding.
   * Jaundice in the past 6 months.
3. - History of drug abuse.
4. - History of renal impairment or severe hepatic impairment.
5. - History or presence of psychiatric disorders
6. - Have donated 500 mL or more blood within 90 days before receiving the first dose of study drug.
7. - Major illness during 3 months before screening.
8. - Subjects who have participated in another clinical study in the past 3 months prior to commencement of this study.
9. - Any difficulty in accessibility of forearm veins for cannulation or blood sampling and or difficulty with donating blood.
10. - Refuse to abstain from food for at least 10 h prior to dosing and for at least 4 h after dosing in each period and for at least 10 h before and at least 4 h after collecting the baseline assessment blood sample in Period 1.
11. - Refuse to abstain from fluid for at least 1 h before and 1 h after dosing.
12. - Refuse to abstain from alcohol for the duration of the study.
13. - Positive during breath alcohol test.
14. - Positive during urine drug screening.
15. - History of difficulty in swallowing study formulations.
16. - Received any medication [including over-the-counter products, vitamins, herbal products] for 14 days preceding the study.
17. - Use of enzyme modifying drugs, MAO inhibitors within 30 days prior to receiving the first dose of study medication.
18. - History of dehydration from diarrhea, vomiting or any other reason within a period of 24 hours prior to study check-in of each period.
19. - Consumption of xanthine containing food and beverages (chocolates, tea, coffee or cola drinks) for at least 48 hours prior to study check-in.
20. - Consumption of grapefruit juice within the 7-days prior to study check-in.
21. - Pregnant females as determined by positive test for pregnancy.
22. - Lactating females.
23. - Investigator/physician feels that it is not in the subject's and/or study's best interest to enroll the subject.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Measurements of pharmacokinetic parameters of each drug | 23 days
  Plasma concentration versus time curves of Dexamethasone and Betamethasone given orally and intramuscularly to non-pregnant females.
Measurements of pharmacodynamic parameters of each drug | 23 days
  Measurements of glucose, cortisol and lymphocyte population changes versus time resulting from the steroid treatment given orally and intramuscularly to non-pregnant females.

SECONDARY OUTCOMES:
Adverse Events | 23 days
  To monitor the adverse events and to ensure the safety of the subjects. Safety assessments will be analyzed descriptively. All continuous variables will be summarized using the following descriptive statistics: n, mean, standard deviation, median, minimum value, and maximum value. Categorical variables will be summarized using frequency counts and percentages. No formal statistical inferences are planned.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Jobe, MD, Ph.D, Study Director — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Syngene International Limited, Tower I, Bangalore, India

IPD SHARING:
Plan to Share IPD: No